CLINICAL TRIAL: NCT02088294
Title: Imagine HEALTH (Healthy Eating Active Living Total Health) Study: Guided Imagery Lifestyle Intervention to Promote Health and Prevent Diabetes in Youth
Brief Title: Guided Imagery Lifestyle Intervention to Promote Health and Prevent Diabetes in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Marc Weigensberg, Associate Professor, Clinical Pediatrics, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NCCAM 1 RO1 AT008330-01
Record Dates: First submitted 2014-02-26; First posted 2014-03-14 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Obesity; Insulin Resistance; Stress
Keywords: obesity; stress; intuitive eating; guided imagery; adolescents; insulin resistance; latinos; minorities
MeSH Terms: conditions — Obesity; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Non-intervention control (No Intervention): No intervention will be delivered.
- Lifestyle Education (LS) (Experimental): The lifestyle curriculum will be taught in twice weekly after-school sessions of ~1.25 hours, one physical activity and one nutrition-related, delivered over 12-weeks during the course of a single academic semester. The lifestyle program will utilize the "Shape Up" curriculum of SOSMentor, a community non-profit collaborator, modified to seamlessly integrate key concepts of the non-diet philosophy of "Intuitive Eating". The curriculum fully encompasses health-promoting nutrition and physical activity practices consistent with consensus recommendations .
  Interventions: Behavioral: Lifestyle Education (LS)
- LS + Stress Reduction Guided Imagery (Experimental): In addition to the after school lifestyle classes, participants will receive group Interactive Guided Imagery (IGI) consisting of standard stress reduction imagery practices, delivered once weekly for 12 weeks as an after school class of ~1.25 hours. The group IGI will be delivered by certified facilitators in the context of the facilitated group process known as "Council", a group communication process used by many indigenous and other cultures.
  Interventions: Behavioral: Lifestyle Education (LS); Behavioral: LS + Stress Reduction Guided Imagery
- LS + Activity/Eating Guided Imagery (Experimental): In addition to the after school lifestyle classes, participants will receive group Interactive Guided ImagerySM (IGI) delivered once weekly for 12 weeks as an after school class of ~1.25 hours. The group IGI will be delivered by certified facilitators in the context of the facilitated group process known as "Council", a group communication process used by many indigenous and other cultures. Participants in this arm will receive stress reduction IGI for 4 wks, plus 8 weekly sessions with IGI content designed to promote physical activity and healthy eating.
  Interventions: Behavioral: Lifestyle Education (LS); Behavioral: LS + Activity/Eating Guided Imagery

INTERVENTIONS:
Behavioral: Lifestyle Education (LS) — See arm description
  Arms: LS + Activity/Eating Guided Imagery; LS + Stress Reduction Guided Imagery; Lifestyle Education (LS)
Behavioral: LS + Stress Reduction Guided Imagery — See Arm Description
  Arms: LS + Stress Reduction Guided Imagery
Behavioral: LS + Activity/Eating Guided Imagery — See arm description
  Arms: LS + Activity/Eating Guided Imagery

SUMMARY:
The childhood obesity epidemic, which falls disproportionately on Latino adolescents, represents a major public health threat to the current generation of youth, and therefore to the health of the nation overall. This project directly addresses the role of psychosocial stress in promoting obesity and metabolic disease risk, and investigates the role of the mind-body CAM intervention of guided imagery in both reducing stress and promoting healthy lifestyle behaviors that could dramatically improve the metabolic health of today's youth.

DETAILED DESCRIPTION:
The childhood obesity epidemic represents a major health threat to the current generation of youth, and falls disproportionately on urban, Latino adolescents. Data suggests modern inner-city minority youth suffer from high levels of psychosocial stress, and that such chronic stress contributes to obesity and insulin resistance, increasing risk of type 2 diabetes, cardiovascular disease, fatty liver disease, and other obesity-related disorders. Guided imagery is a mind-body complementary/alternative medicine (CAM) modality that offers promise as a therapeutic intervention to reduce psychosocial stress, and also to promote healthy lifestyle behaviors. In a pilot 12-week lifestyle intervention, Interactive Guided ImagerySM significantly reduced salivary cortisol, reduced sedentary behavior, and increased moderate physical activity in overweight Latino adolescents. The overall aim of this proposal is to determine the separate contributions of stress reduction guided imagery and health behavior guided imagery, when delivered in the context of a health-promoting, lifestyle intervention, on short-term and long-term stress-reduction and behavioral outcomes in predominantly Latino high school students. The study consists of a high school-based, 12-week lifestyle intervention delivered in an after school program to urban, predominantly Latino adolescents. The intervention features a health-promoting, lifestyle education class, combined with a group guided imagery intervention that is theoretically grounded in Self-Determination Theory (SDT). High school students are randomized to one of 4 intervention arms 1) Non-intervention control; 2) lifestyle education alone (LS); 3) LS + Stress Reduction guided imagery alone; 4) LS + Physical Activity/Healthy Eating guided imagery. Outcomes will be measured upon completion of the 12-wk intervention, after an additional 6-month maintenance program, and after a further 6-month period of no program contact. Primary outcomes will be change in salivary cortisol patterns and changes in physical activity and dietary intake. Secondary outcomes are insulin resistance, body fat, carotid intima media thickness, metabolic syndrome, perceived stress, well-being (self-esteem, health related quality of life), and measures of mediation by SDT constructs. Results will demonstrate the isolated effects of the lifestyle education and the two different forms of guided imagery, and could shift the paradigm of obesity prevention and treatment in urban minority youth to include attention to social stress and promotion of well-being.

ELIGIBILITY:
Inclusion Criteria:

* Male and female enrolled in second year (i.e. sophomore year) of high school at time of consent into study, junior year at time of intervention
* Self-stated intent to complete high school
* Predominantly minority ethnicity (self-reported)
* Overweight/ obese and normal weight
* Agreement to attend up to 3 after school classes per week for the 12 weeks of the program

Exclusion Criteria:

* Serious chronic illness or physical, cognitive, or behavioral disability that would prevent ability to fully receive intervention
* Prior diagnosis of clinical eating disorder, psychiatric disorder, or significant cognitive disability
* Lack of English fluency
* Participation in previous "Council" programs offered through the school
* Participation in formal weight-loss programs in 3 months preceding entry to study
* Pregnancy
* Sibling or other household member enrolling for the intervention

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Physical activity | 3 months
  Physical activity and sedentary behavior will be measured by accelerometry and 3-day physical activity recall.

SECONDARY OUTCOMES:
Change in Salivary Cortisol, daily slope | 3 months
  Salivary cortisol will be collected on 3 successive days at awakening, 30-minutes post-awakening, and in the evening.
Change in Dietary intake | 3 months
  Dietary intake of macronutrients measured by 3-day diet record

OTHER OUTCOMES:
Change in Perceived Stress | 3 months
  Measured by Perceived Stress Scale
Change in Well-Being | 3 months
  Measured by Psychological General Well-Being Index (GWBS) and the Arizona Integrated Outcomes Scale.
Change in Adiposity | 3 months
  BMI will be determined based on standards for age and sex, using clinical balance and stadiometer. Percent body fat will be determined by bioimpedance.
Change in Insulin resistance | 3 months
  The Homeostatic Model Insulin Resistance Index will be determined based on measures of fasting glucose and insulin.
Change in Carotid artery intima media thickness | 15 months
  Determined by carotid artery ultrasound.
Change in Self-determination Theory Constructs | 3 months
  Constructs of SDT will be assessed as theoretical mediators of intervention effects using the following survey measures: Perceived Competence for Participating in Regular Physical Activity (PCSPA) and for Healthy Eating (PCSHE); Health Care Climate Questionaire to determine autonomy support; Exercise Self-Regulation Questionnaire and Treatment Self-Regulation Questionnaire to determine autonomous motivation for physical activity and healthy eating; Group Cohesion Scale to assess relatedness.
Change in Intuitive eating | 3 months
  Intuitive Eating Scale measures attitudes and behaviors relating to intuitive eating.

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Weigensberg, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Derived] Toledo-Corral CM, Ding L, Morales JC, Chapman TM, Romero MB, Weigensberg MJ. Morning Serum Cortisol Is Uniquely Associated with Cardiometabolic Risk Independent of Body Composition in Latino Adolescents. Metab Syndr Relat Disord. 2023 May;21(4):214-221. doi: 10.1089/met.2022.0091. Epub 2023 Apr 11. PMID 37042653
- [Derived] Sumner JA, Gao X, Gambazza S, Dye CK, Colich NL, Baccarelli AA, Uddin M, McLaughlin KA. Stressful life events and accelerated biological aging over time in youths. Psychoneuroendocrinology. 2023 May;151:106058. doi: 10.1016/j.psyneuen.2023.106058. Epub 2023 Feb 17. PMID 36827906
- [Derived] Bell BM, Spruijt-Metz D, Naya CH, Lane CJ, Wen CKF, Davis JN, Weigensberg MJ. The mediating role of emotional eating in the relationship between perceived stress and dietary intake quality in Hispanic/Latino adolescents. Eat Behav. 2021 Aug;42:101537. doi: 10.1016/j.eatbeh.2021.101537. Epub 2021 Jun 30. PMID 34225165
- [Derived] Weigensberg MJ, Avila Q, Spruijt-Metz D, Davis JN, Wen CKF, Goodman K, Perdomo M, Wade NB, Ding L, Lane CJ. Imagine HEALTH: Randomized Controlled Trial of a Guided Imagery Lifestyle Intervention to Improve Obesity-Related Lifestyle Behaviors in Predominantly Latinx Adolescents. J Altern Complement Med. 2021 Sep;27(9):738-749. doi: 10.1089/acm.2020.0515. Epub 2021 May 25. PMID 34037459
- [Derived] Weigensberg MJ, Spruijt-Metz D, Wen CKF, Davis JN, Avila Q, Juarez M, Brown-Wade N, Lane CJ. Protocol for the Imagine HEALTH Study: Guided imagery lifestyle intervention to improve obesity-related behaviors and salivary cortisol patterns in predominantly Latino adolescents. Contemp Clin Trials. 2018 Sep;72:103-116. doi: 10.1016/j.cct.2018.07.009. Epub 2018 Aug 2. PMID 30076988